CLINICAL TRIAL: NCT00181844
Title: A Pilot Open Study of the Safety and Effectiveness of Lamotrigine for the Treatment of Mania in Youth Ages 6-17 With Bipolar I, Bipolar II, and Bipolar Spectrum Disorders
Brief Title: Lamotrigine for the Treatment of Mania in Youth Ages 6-17 With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Assistant Professor of Psychiatry at Harvard Medical School and at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-P-001419
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-03

CONDITIONS: Bipolar Disorder; Mania
Keywords: bipolar disorder; lamotrigine; children; mania
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lamotrigine (Experimental)
  Interventions: Drug: lamotrigine

INTERVENTIONS:
Drug: lamotrigine — Open-label, flexible-dose, BID treatment of lamotrigine (Lamictal). For children <12 years, dosing began at 0.35 mg/kg/day, divided in 2 doses, rounded down to nearest 5mg, to be increased weekly depending on response and tolerability to maintenance dose of 5-15 mg/kg/day (maximum 400 mg/day in 2 divided doses). For children ≥12 years, dose began at 25 mg/day in 1 dose, to be increased weekly depending on response and tolerability to maintenance dose of 300-500 mg/day in 2 divided doses.
  Other Names: Lamictal

SUMMARY:
The main objective of this study is to assess the effectiveness and safety of lamotrigine in the treatment of youth with bipolar and bipolar spectrum disorder. This is an exploratory, 12-week, open-label treatment period, pilot study, of youth ages 6-17, who meet the DSM-IV diagnostic criteria for bipolar I, bipolar II, or bipolar spectrum disorder. The study results will be used to generate hypotheses for a larger randomized controlled clinical trial. Based on the available literature in adults with bipolar disorder, we hypothesized that lamotrigine will be efficacious and well tolerated in youth with pediatric bipolar and bipolar spectrum disorders.

DETAILED DESCRIPTION:
Lamotrigine is a new generation antiepileptic drug, approved by the FDA in 2003 for the maintenance treatment of adults with Bipolar I disorder to delay the time to occurrence of mood episodes (depression, mania, hypomania,& mixed episodes) in patients treated for acute mood episodes with standard therapy. Recent studies have shown that Lamotrigine maintenance treatment was more robust in bipolar depression.

The study includes 1) use of a 12-week design to document the response rate 2) assessment of the impact of Lamotrigine on functional capacities and cognition, 3) careful assessment of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 6-17 years of age.
2. Subjects must have a DSM-IV diagnosis of bipolar I, bipolar II disorder or bipolar spectrum disorder and currently displaying manic, hypomanic, or mixed symptoms (with or without psychotic features) according to the DSM-IV based on clinical assessment and confirmed by structured diagnostic interview (Kiddie Schedule of Affective Disorders and Schizophrenia Epidemiological Version. Bipolar Spectrum Disorder (or sub-threshold bipolar disorder) is operationalized as having severe mood disturbance, which meets DSM-IV Criteria A for bipolar disorder but meet fewer elements in criteria B (only require 2 items for elation category and 3 for irritability).
3. Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
4. Subjects and their legal representative must be considered reliable.
5. Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.
6. Subjects must have an initial score on the Y-MRS total score of at least 20.
7. Subject must be able to participate in mandatory blood draws.
8. Subject must be able to swallow pills.
9. Subjects with comorbid ADHD, ODD, CD, anxiety and depressive disorders will be allowed to participate in the study provided they do not meet for any of the exclusionary criteria.
10. For concomitant stimulant therapy used to treat ADHD, subjects must have been on a stable dose of the medication for 1 month prior to study enrollment. The dose of the stimulant therapy will not change throughout the duration of the study.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Subjects unable to swallow pills.
3. Serious, unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
4. History of sensitivity to lamotrigine or known, severe allergies or multiple adverse drug reactions.
5. History of previous bone marrow depression.
6. History of serious rashes.
7. DSM-IV substance (except nicotine or caffeine) dependence within past 3 months.
8. Judged clinically to be at serious suicidal risk.
9. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol.
10. A non-responder or a history of intolerance to lamotrigine in an adequate trial (2 months or more at an adequate dose) as determined by the clinician.
11. Current diagnosis of schizophrenia.
12. Pregnant or nursing females.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2005-01; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Signed Consent
Arm/Group | Lamotrigine
Started | 51
Completed | 39
Not Completed | 12
Not completed — Withdrawal by Subject | 5
Not completed — Did not meet entrance criteria | 7
Period: Exposed to Study Medication
Arm/Group | Lamotrigine
Started | 39
Completed | 22
Not Completed | 17
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 2
Not completed — Non-compliance | 2
Not completed — Withdrawal by Subject | 1
Not completed — Difficulty meeting study schedule | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lamotrigine
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Change of Mania Symptoms Assessed by Young Mania Rating Scale (YMRS)
Description: Mean reduction in YMRS score at endpoint/LOCF. This is a scale to measure symptoms of mania in children and adolescents. 11 items are rated from 0-4 (7 items) or 0-8 (4 items). The minimum (least severe) total score is 0, and maximum (most severe) total score is 60.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 39
Units on a scale | -14.9 (9.7)

ADVERSE EVENTS:
Arm/Group | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 34/39
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamotrigine (N=39)
Acid reflux (Gastrointestinal disorders) | 1 (5)
Appetite loss (Gastrointestinal disorders) | 3 (4)
Backache (General disorders) | 1 (1)
Bruising (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Cold (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Ear and labyrinth disorders) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (5)
Ear infection (Infections and infestations) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 3 (4)
Eye irritation (Eye disorders) | 2 (2)
Fatigue (General disorders) | 5 (9)
Fever (General disorders) | 5 (6)
GERD vomiting (Gastrointestinal disorders) | 1 (2)
Headache (General disorders) | 15 (37)
Hip dysplasia (Musculoskeletal and connective tissue disorders) | 2 (2)
Increased appetite (General disorders) | 1 (2)
Injury (Injury, poisoning and procedural complications) | 11 (17)
Insomnia (General disorders) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 3 (3)
Jitteriness (General disorders) | 2 (2)
Lethargy (General disorders) | 2 (8)
Loss of voluntary movement (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Menstrual cramps (Reproductive system and breast disorders) | 1 (1)
More manic (Psychiatric disorders) | 1 (1)
Nasal congestion (General disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 4 (10)
Nosebleed (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Panic attacks (Psychiatric disorders) | 2 (4)
Poison Ivy (Injury, poisoning and procedural complications) | 1 (1)
Rhinorhea (General disorders) | 4 (5)
Shakiness (General disorders) | 2 (2)
Sinus infection (Infections and infestations) | 1 (1)
Sore throat (General disorders) | 7 (8)
Stomach ache (Gastrointestinal disorders) | 7 (15)
Temper tantrum (General disorders) | 2 (2)
Tooth pain (General disorders) | 6 (8)
Unsteady (General disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (13)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rashes (Skin and subcutaneous tissue disorders) | 7
Contact dermatitis (Skin and subcutaneous tissue disorders) | 2
Sunburn (Skin and subcutaneous tissue disorders) | 2
Miscellaneous other skin lesions (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes